CLINICAL TRIAL: NCT06161597
Title: Family Check-Up Online for Middle School Parents
Brief Title: Family Check-Up Online
Acronym: FCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Arizona Health Care Cost Containment System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00017956
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Families of Middle School Students at Title 1 Schools

STUDY DESIGN:
Intervention Model Description: All participants will receive the primary intervention: The Family Check-Up Online. Participants will then be randomly assigned to a specific coaching condition.
Masking Description: Study personnel and participants are informed of what condition participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informational Support (Experimental): Parents will be told that they have the option of contacting an informational support specialist any point while completing the program to address questions and discuss the program. Parents will be informed that their questions can be addressed via e-mail or alternatively they can schedule a time to talk with their coach via phone or Zoom. The informational support specialist will not initiate contact with parents in this condition.
  Interventions: Behavioral: Family Check-Up Online
- Guidance Coaching (Experimental): Parents will be informed that they have been assigned a guidance coach who will contact them via email to schedule 1-3 check-in meetings over the phone or via Zoom while they complete the online program. These meetings are structured to help establish parental goals for the program, offer emotional support, and help motivate parents to implement new parenting skills. During these contacts, coaches use motivational interviewing techniques to help promote and support behavioral change. These coaching contacts are designed to be brief and focused, and typically last for less than 30 minutes. Coach contacts are scheduled based on the parents' availability and interest, and additional coaching sessions can be requested by the parent at any point during the program.
  Interventions: Behavioral: Family Check-Up Online

INTERVENTIONS:
Behavioral: Family Check-Up Online — Families will be provided with access to the FCO program, available in English or Spanish. Parents complete a tutorial and five different modules focused on distinct parenting skills. Each module starts with a survey and feedback to help identify relative strengths and challenges with the targeted parenting skills. Parents are then guided through various online activities including videos that model right and wrong ways to handle comm on situations and explanations of parental self-management and problem-solving strategies. Parents are complete activities to practice the parenting skills taught. Parents will have access to the online program for 8 and they are encouraged to practice the program strategies during this time period. At the end of the 8 weeks, parent re-complete the brief questions that they filled out at the beginning of each module and then receive feedback indicating which of the parent's domain scores have improved since they completed each module.

SUMMARY:
The goal of this clinical trial is to test the benefits of the Family Check-Up Online Program for parents of middle school students in Arizona. Participants will complete an online pre-survey, gain access to the online parenting program Family Check-Up, and have the option to meet with a coach to discuss the program. The participants will also complete a post-survey 3 months after enrollment.

DETAILED DESCRIPTION:
The lingering impact of the COVID-19 pandemic has impacted families adversely in multiple ways, including economic stressors, mental health-related functioning, and social/familial functioning. Given the scale of the pandemic's impact on families with school-aged children, the implementation of effective family-focused programs that target core mechanisms of change with a broad range of benefits for parents and youth across diverse populations, and that can be brought to scale rapidly and with fidelity, represents critical public health goals.

Toward this end, this project is designed to further examine the efficacy of a web-based version of the universal Family Check-Up prevention program, which is an empirically-supported, parent-focused program designed to promote resilience and improve family functioning among parents of middle school-aged youth (grades 6-8th). A randomized control trial conducted through the University of Oregon found that parents who completed the Family Check-up Online program (FCO) either with or without supplemental support coaching exhibited significant increases in confidence and effortful control related to implementing skills and strategies that promote positive emotional and behavioral health among teens. This suggests that parents who complete the program feel more empowered to help guide their child's positive decision making and more effectively manage family challenges.

This project will examine whether the FCO program produces improvements in positive parenting practices, reductions in parental emotional distress, and reductions in youth emotional/behavioral problems when delivered as a universal prevention program targeting parents of 6-8th grade students attending Title 1 public schools (>50% students eligible for free/reduced lunch). The investigators will also examine whether the structured parent coaching support component of the program (i.e., Guidance Coaching) helps to improve the program's effectiveness relative to a parent-initiated informational support condition.

ELIGIBILITY:
Inclusion Criteria:

* All parents with a child enrolled in grades 6-8 at participating Title 1 public schools will be invited to take part in the study.

Exclusion Criteria:

* N/A

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Active Parental Monitoring | 3 months
  Parent self-report of monitoring, range 1-5, higher values = better outcome
Positive Parenting | 3 months
  Parent self-report of positive parenting practices, range 1-5, higher values = better outcome
Harsh Parenting | 3 months
  Parent self-report of harsh parenting, range 1-5, higher values = worse outcome
Parental Confidence | 3 months
  Parent self-report of confidence with various parenting strategies, range 1-5, higher values = better outcome
Child Anger | 3 months
  Parent report of their child's anger, range 1-5, higher values = worse outcome
Child Oppositional Defiance | 3 months
  Parent report of their child's oppositional defiant behavior, range 1-5, higher values = worse outcome
Child Callous-Unemotional Traits | 3 months
  Parent report of their child's callousness, range 1-5, higher values = worse outcome
Child Aggression | 3 months
  Parent report of their child's aggression, range 1-5, higher values = worse outcome
Child School Performance | 3 months
  Parent report of their child's school performance, range 1-5, higher values = better outcome
Child Stress | 3 months
  Parent report of child's stress with PROMIS scale, range 1-5, higher values = worse outcome
Child Anxiety | 3 months
  Parent report of child's anxiety with PROMIS scale, range 1-5, higher values = worse outcome
Child Depression | 3 months
  Parent report of child's depression with PROMIS scale, range 1-5, higher values = worse outcome
Family Conflict | 3 months
  Parent report of family conflict including arguing and fighting, range 1-5, higher values = worse outcomes

SECONDARY OUTCOMES:
Parent Anxiety | 3 months
  Parent self-report of anxiety with PROMIS scale, range 1-5, higher values = worse outcome
Parent Depression | 3 months
  Parent self-report of depression with PROMIS scale, range 1-5, higher values = worse outcome
Parent Stress | 3 months
  Parent self-report of stress with PROMIS scale, range 1-5, higher values = worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT06161597/ICF_000.pdf